CLINICAL TRIAL: NCT04362540
Title: Is Fat in the Liver a Marker of Post-Pregnancy Glycaemic Deterioration in Women With Gestational Diabetes?
Acronym: FLiP-GD2
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor
Other Study IDs: 214643
Record Dates: First submitted 2020-02-14; First posted 2020-04-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Magnetic Resonance Imaging; Glucose Tolerance Test; Ultrasonography; Metabolome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with GDM: Ultrasound liver scan in addition to routine foetal assessment (antenatal) Metabolic profile blood tests, Oral Glucose Tolerance Test, ELF blood test, repeat liver ultrasound scan and MRI scan (post partum)
  Interventions: Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: MRI scan — On attendance to antenatal clinic with confirmed diagnosis of gestational diabetes based on OGTT and following informed consent: Ultrasound scan: Those with positive OGTT results (i.e. GDM positive) will attend an appointment for an ultrasound scan, as per routine practice. These women will,at that appointment, be assessed for presence/absence of NAFLD as well as undergoing their routine foetal assessment. This is a simple addendum to the existing scan, taking no more than 5 minutes. Participants will have been informed during the consent process that the results (regarding the presence / absence of NAFLD) will be compared to MRI after delivery.
  Other Names: OGTT; ELF; Ultrasound; Metabolic Profile

SUMMARY:
The aim of this study is to utilise ultrasound, using an established method for detecting NAFLD, to determine whether the presence of NAFLD in women with GDM, detected during routine scanning, is a marker of deterioration in glycaemic status post-partum. We propose to assess the relationship between NAFLD and surrogates for insulin resistance as well as glycaemic status, insulin sensitivity and β-cell function, after delivery.

The study is not seeking to compare the incidence of T2DM between those with and without NAFLD. This would require a longer follow-up and larger cohort size. Instead, it aims to quantify the degree of early deterioration of glycaemic status in these groups using insulin resistance markers. This is a clinically important issue as a greater level of insulin resistance would in itself trigger clinical intervention, including vigilant follow-up and empowerment for proactive healthy life style changes, which have been shown to prevent diabetes development .

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Pregnant women diagnosed with GDM based on OGTT

Exclusion Criteria:

* Women with known type 1 or type 2 diabetes prior to pregnancy
* Women with known history of liver disease including alcoholic liver disease
* Women unable or unwilling to consent to be part of the study
* Women with contraindication to MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with GDM as defined in routine practice, using standard oral glucose tolerance testing (OGTT). Women with confirmed GDM will be classified as either NAFLD-positive or NAFLD-negative on the basis of postpartum MRI scan.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure for the study will be the mean difference in values of the HOMA-IR (as a surrogate for insulin resistance) in those with NAFLD vs. those without NAFLD 6-12 weeks post partum | 6-12 weeks post partum
  To determine whether the presence of NAFLD during pregnancy in women with gestational diabetes mellitus is a marker of worse metabolic profile (insulin resistance).

SECONDARY OUTCOMES:
Comparison of HbA1c and fasting glucose (standard markers of dysglycaemia) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of disposition index (marker of insulin resistance) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of QUICKI (marker of insulin resistance) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of insulin and nonesterified fatty acid levels (marker of insulin resistance) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of fasting levels from a 4 point OGTT (marker of insulin resistance) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of area-under-the-curve from 4 point OGTT (marker of insulin resistance) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of ELF blood test results (advanced marker of insulin resistance) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of liver function tests (as part of the Fatty Liver Index) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of Body Mass Index (as part of the Fatty Liver Index) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of waist circumference (as part of the Fatty Liver Index) in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
Comparison of alcohol history in those with NAFLD vs. those without NAFLD at 6-12 weeks post partum | 6-12 weeks post partum
The presence of fat in the liver using a liver ultrasound scan at baseline and 6-12 weeks post partum. | 6-12 weeks post partum
MRI scan to confirm the presence of NAFLD at 6-12 weeks post partum. | 6-12 weeks post partum

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No